CLINICAL TRIAL: NCT05674500
Title: A Prospective Study of Standardized Coaching Language to Improve Endoscopy Training Quality
Brief Title: Coaching Language to Improve Endoscopy Training Quality
Acronym: CLIEnT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Roopa Vemulapalli, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU-2021-0829
Record Dates: First submitted 2022-12-09; First posted 2023-01-06 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Education, Medical; Colonoscopy
Keywords: Faculty; Fellows; Simulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Faculty participants will participate in educational training designed to teach them standardized coaching language for endoscopy instruction and strategies to promote effective communication during an endoscopy teaching. It will be comprised of:
  1. A 15-minute-long training video demonstrating the use of recommended coaching language for endoscopy instruction (e.g., recommended 14 standard terms, need to refer to the screen when directing a trainee as opposed to their hands, use of a clockface analogy) and communication best practices (e.g., checking to ensure understanding, avoidance of cognitive overload, task deconstruction)
  2. The faculty will be given a small (10x10 cm) flash card with the recommended 14 standard terms which they can access during the second simulated encounter. To control for any potential effect of the presence of the card on the trainee during teaching, each faculty be given an identical card with 14 random words on it to hold during the first encounter
  Interventions: Other: Educational Training on standardized coaching language
- Control Group (Active Comparator): Faculty participants will take part in 'dummy' educational training comprised of:
  1. A 15-minute-long 'dummy' colonoscopy training video which outlines how to set goals ahead of an endoscopy training session. The video will not discuss standardized coaching language and/or communication best practices
  2. This group will also be provided a small (10x10cm) flash card but with random words on it (identical to the first simulated colonoscopy teaching encounter).
  Interventions: Other: Educational Training on goal setting

INTERVENTIONS:
Other: Educational Training on standardized coaching language — The faculty trainer participants in training groups will watch a 15-min long video between the two simulated endoscopy teaching encounters. The video link will be emailed to them 1 week before the second simulated encounter, and they can watch it in their own time. The training video will demonstrate the use of recommended coaching language for endoscopy instruction (e.g., recommended 14 standard terms, need to refer to the screen when directing a trainee as opposed to their hands, use of a clockface analogy) and communication best practices (e.g., checking to ensure understanding, avoidance of cognitive overload, task deconstruction).
  Arms: Training Group
Other: Educational Training on goal setting — The faculty trainer participants in the control groups will watch a 15-min long video between the two simulated endoscopy teaching encounters. The video link will be emailed to them 1 week before the second simulated encounter, and they can watch it in their own time. The video will be a 'dummy' colonoscopy training video which outlines how to set goals ahead of an endoscopy training session. The video will not discuss standardized coaching language and/or communication best practices.
  Arms: Control Group

SUMMARY:
The goal of this randomized control study is to determine if the use of standardized coaching language by faculty trainers for teaching colonoscopy is associated with improved colonoscopy performance. The main questions it aims to answer are:

* If the use of standardized coaching language is effective in improving colonoscopy training?
* If the use of standardized coaching language influences the clarity of instructions by the faculty trainers during colonoscopy teaching Participants will take part in simulated colonoscopy teaching encounter using a virtual reality simulator for 1 hour in 2 different sessions 2 weeks apart.

Researchers will compare 2 groups of faculty trainers to to see if the standardized coaching language effects the colonoscopy training quality.

ELIGIBILITY:
Inclusion Criteria:

* Faculty members who are endoscopy trainers in either pediatric or adult gastroenterology division at University of Texas Southwestern Medical Center or Children's Medical Center, Dallas
* Fellow trainees in pediatric or adult gastroenterology division at University of Texas Southwestern Medical Center or Children's Medical Center, Dallas

Exclusion Criteria:

* Advanced endoscopy fellows
* Fellows beyond Post-Graduate Year-6 (PGY-6)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in colonoscopy performance | Change from Baseline colonoscopy performance at 2 weeks
  The de-identified video-recording of the simulated colonoscopy will be assessed by blinded external rater.
  This will be done using the Gastrointestinal Endoscopy Competency Assessment Tool (GiECAT) which is a colonoscopy assessment tool with strong validity evidence. For the GiECAT, 6 global rating items on supervision scale (measuring from 1 to 5) and 5 checklist items which are applicable to simulated procedures (i.e., no patients involved) will be used. Since it is a competency based tool with a checklist, there is no maximum score, but instead is a rating scale.
  To ensure blinding, only the trainee's gloved hands will be seen, and the videos used for assessment of colonoscopy performance will not have sound to control for any effects the faculty instruction may have on the ratings of performance.
Change in colonoscopy performance | Change from Baseline colonoscopy performance at 2 weeks
  The de-identified video-recording of the simulated colonoscopy will be assessed by blinded external rater.
  This will be done using another colonoscopy assessment form with strong validity evidence - 8 'Procedure' items from the Joint Advisory Group on GI Endoscopy (JAG) Colonoscopy Direct Observation of Procedural Skills (DOPS) form. This is a supervision-based scale (measuring from 1 to 4). Since this is also a competency based tool with a checklist, it has a rating scale with no maximum score.
  To ensure blinding, only the trainee's gloved hands will be seen, and the videos used for assessment of colonoscopy performance will not have sound to control for any effects the faculty instruction may have on the ratings of performance.

SECONDARY OUTCOMES:
Change in 'Red-out' time | Change from baseline time in red-out at 2 weeks
  The percentage of procedure time during which the endoscope tip (camera) was against the mucosa of the virtual bowel (i.e., there was no proper visualization of the bowel mucosa - appears as 'reddened out screen', aka 'red-out'), as auto-generated automatically by the colonoscopy simulator. The percentage ranges from 0 to 100.
Change in time to cecum | Change from baseline time to cecum at 2 weeks
  The time it took the trainee to reach the cecum, as auto-generated automatically by the colonoscopy simulator. This is reported in minutes and seconds (min:sec). The range from 0 to 20 minutes
Change in Cognitive load | Change from Baseline cognitive load at 2 weeks
  Printed forms will be given to all participants immediately after the pre-and post-sessions to measure the cognitive load. It will be measured by 3 measurement tools (Outcome 5-7) Overall cognitive load: A single item rating tool asking participants to rate the amount of mental effort they required to complete the simulated endoscopy on a 9-point scale (1 = very, very small effort and 9 = very, very high effort).
Change in Cognitive load | Change from Baseline cognitive load at 2 weeks
  Printed forms will be given to all participants immediately after the pre-and post-sessions to measure the cognitive load.
  NASA Task Load Index (NASA-TLX): A 6-item rating scale with strong validity evidence that assesses perceived demand, effort and frustration in performing the task, with higher scores indicating an increased cognitive load (Ranges from 0 to 20).
Change in Cognitive load | Change from Baseline cognitive load at 2 weeks
  Printed forms will be given to all participants immediately after the pre-and post-sessions to measure the cognitive load.
  Cognitive Load Index for Colonoscopy (for trainees ONLY): A measure of intrinsic, extraneous, and germane cognitive load related to performing colonoscopy. Fifteen items that are applicable to the simulation will be rated. Given the nature of this scale, it will be administered to trainees only. Scale ranges from 1 (strongly disagree) to 10 (strongly agree).
Change in the Clarity of instruction (trainee's perception) | Change from Baseline trainer's language assessment at 2 weeks
  The clarity of instruction will be rated by the trainee on a Likert scale, using linguistics specific metrics developed an expert in linguistics. Description-based scale with following categories- Excellent, Satisfactory, Needs Improvement and Not Acceptable.
  This form will be provided to the trainees only to assess their perception of the instructions provided by the faculty instructor.
Change in the trainer's language (assessed by linguistics expert) | Change from Baseline trainer's language assessment at 2 weeks
  Based on the de-identified video recordings, the trainer's clarity of instructions and use of recommended language will be rated using specialized linguistic-designed assessment rubric by a blinded external linguistics expert.
  Name of Measurement- Clarity of language and use of standardized terminology Measurement Tool- Linguistics rubric (descriptive rating scale, with following categories- Excellent, Satisfactory, Needs Improvement and Not Acceptable)
Semi-structured interview of the trainees | At 2 weeks
  In order to complement and enhance the data from above mentioned assessment tools (i.e., clarity of instruction, cognitive load), trainees will be asked to participate in a short 10-15 minute interview with the PI and/or Co-PI after the they have completed all 4 simulated cases, to explore their perceptions of instruction provided. The interview guide has been adapted from a study examining gastroenterology trainees' perception of endoscopy training activities. Interviews will be transcribed (removing any identifiers) and coded qualitatively using a constant comparison approach to compare differences in trainee's perceptions between groups
Semi-structured interview of the faculty instructor | At 2 weeks
  In order to explore faculty's perceptions of the training modality being tested, faculty participants will also be asked to participate in a separate 10-15 minute long semi-structured interview with the PI and/or co-PI, after completing the 2 simulation sessions with a trainee fellow. The interview guide has been adapted from a study exploring endoscopy trainers' experience in teaching endoscopy. Interview will be transcribed and coded qualitatively using a constant comparison approach to explore the faculty's perception of the instructional strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Aayush Gabrani, MD, Principal Investigator — University of Texas
Locations (1):
- UTSW, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared because this was not included in the consent form at the time of study design. Most of the participants have already been consented and recruited to participate and IPD was not included in that discussion.

REFERENCES:
- [Background] Walsh CM. In-training gastrointestinal endoscopy competency assessment tools: Types of tools, validation and impact. Best Pract Res Clin Gastroenterol. 2016 Jun;30(3):357-74. doi: 10.1016/j.bpg.2016.04.001. Epub 2016 Apr 16. PMID 27345645
- [Background] Waschke KA, Anderson J, Macintosh D, Valori RM. Training the gastrointestinal endoscopy trainer. Best Pract Res Clin Gastroenterol. 2016 Jun;30(3):409-19. doi: 10.1016/j.bpg.2016.05.001. Epub 2016 May 14. PMID 27345649
- [Background] Siau K, Green JT, Hawkes ND, Broughton R, Feeney M, Dunckley P, Barton JR, Stebbing J, Thomas-Gibson S. Impact of the Joint Advisory Group on Gastrointestinal Endoscopy (JAG) on endoscopy services in the UK and beyond. Frontline Gastroenterol. 2019 Apr;10(2):93-106. doi: 10.1136/flgastro-2018-100969. Epub 2018 Nov 13. PMID 31210174
- [Background] Coderre S, Anderson J, Rostom A, McLaughlin K. Training the endoscopy trainer: from general principles to specific concepts. Can J Gastroenterol. 2010 Dec;24(12):700-4. doi: 10.1155/2010/493578. PMID 21165376
- [Background] Walsh CM, Anderson JT, Fishman DS. Evidence-based Approach to Training Pediatric Gastrointestinal Endoscopy Trainers. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):501-504. doi: 10.1097/MPG.0000000000001473. PMID 27846065
- [Background] Gavin DR, Valori RM, Anderson JT, Donnelly MT, Williams JG, Swarbrick ET. The national colonoscopy audit: a nationwide assessment of the quality and safety of colonoscopy in the UK. Gut. 2013 Feb;62(2):242-9. doi: 10.1136/gutjnl-2011-301848. Epub 2012 Jun 1. PMID 22661458
- [Background] Broekaert I, Tzivinikos C, Narula P, Antunes H, Dias JA, van der Doef H, Isoldi S, Norsa L, Romano C, Scheers I, Silbermintz A, Tavares M, Torroni F, Urs A, Thomson M. European Society for Paediatric Gastroenterology, Hepatology and Nutrition Position Paper on Training in Paediatric Endoscopy. J Pediatr Gastroenterol Nutr. 2020 Jan;70(1):127-140. doi: 10.1097/MPG.0000000000002496. No abstract available. PMID 31799965
- [Background] Dilly CK, Sewell JL. How to Give Feedback During Endoscopy Training. Gastroenterology. 2017 Sep;153(3):632-636. doi: 10.1053/j.gastro.2017.07.023. Epub 2017 Jul 27. No abstract available. PMID 28757268
- [Background] Zawadzki M, Gomez Ruiz M, Tou S, Jeffels A, Matzel KE. A proposed system for standardized terminology in minimally invasive surgery - a video vignette. Colorectal Dis. 2020 Dec;22(12):2346-2347. doi: 10.1111/codi.15309. Epub 2020 Sep 16. No abstract available. PMID 32790087
- [Background] Lauridsen KG, Watanabe I, Lofgren B, Cheng A, Duval-Arnould J, Hunt EA, Good GL, Niles D, Berg RA, Nishisaki A, Nadkarni VM. Standardising communication to improve in-hospital cardiopulmonary resuscitation. Resuscitation. 2020 Feb 1;147:73-80. doi: 10.1016/j.resuscitation.2019.12.013. Epub 2019 Dec 28. PMID 31891790
- [Background] Khan R, Zheng E, Wani SB, Scaffidi MA, Jeyalingam T, Gimpaya N, Anderson JT, Grover SC, McCreath G, Walsh CM. Colonoscopy competence assessment tools: a systematic review of validity evidence. Endoscopy. 2021 Dec;53(12):1235-1245. doi: 10.1055/a-1352-7293. Epub 2021 Mar 16. PMID 33440438
- [Background] Barton JR, Corbett S, van der Vleuten CP; English Bowel Cancer Screening Programme; UK Joint Advisory Group for Gastrointestinal Endoscopy. The validity and reliability of a Direct Observation of Procedural Skills assessment tool: assessing colonoscopic skills of senior endoscopists. Gastrointest Endosc. 2012 Mar;75(3):591-7. doi: 10.1016/j.gie.2011.09.053. Epub 2012 Jan 9. PMID 22227035
- [Background] Siau K, Dunckley P, Valori R, Feeney M, Hawkes ND, Anderson JT, Beales ILP, Wells C, Thomas-Gibson S, Johnson G; Joint Advisory Group on Gastrointestinal Endoscopy (JAG). Changes in scoring of Direct Observation of Procedural Skills (DOPS) forms and the impact on competence assessment. Endoscopy. 2018 Aug;50(8):770-778. doi: 10.1055/a-0576-6667. Epub 2018 Apr 3. PMID 29614526
- [Background] Siau K, Crossley J, Dunckley P, Johnson G, Feeney M, Iacucci M, Anderson JT; Joint Advisory Group on Gastrointestinal Endoscopy (JAG). Colonoscopy Direct Observation of Procedural Skills Assessment Tool for Evaluating Competency Development During Training. Am J Gastroenterol. 2020 Feb;115(2):234-243. doi: 10.14309/ajg.0000000000000426. PMID 31738285
- [Background] Walsh CM, Ling SC, Khanna N, Grover SC, Yu JJ, Cooper MA, Yong E, Nguyen GC, May G, Walters TD, Reznick R, Rabeneck L, Carnahan H. Gastrointestinal Endoscopy Competency Assessment Tool: reliability and validity evidence. Gastrointest Endosc. 2015;81(6):1417-1424.e2. doi: 10.1016/j.gie.2014.11.030. Epub 2015 Mar 7. PMID 25753836
- [Background] Walsh CM, Ling SC, Mamula P, Lightdale JR, Walters TD, Yu JJ, Carnahan H. The gastrointestinal endoscopy competency assessment tool for pediatric colonoscopy. J Pediatr Gastroenterol Nutr. 2015 Apr;60(4):474-80. doi: 10.1097/MPG.0000000000000686. PMID 25564819
- [Background] Sewell JL, Boscardin CK, Young JQ, Ten Cate O, O'Sullivan PS. Measuring cognitive load during procedural skills training with colonoscopy as an exemplar. Med Educ. 2016 Jun;50(6):682-92. doi: 10.1111/medu.12965. PMID 27170086
- [Background] Sewell JL, Young JQ, Boscardin CK, Ten Cate O, O'Sullivan PS. Trainee perception of cognitive load during observed faculty staff teaching of procedural skills. Med Educ. 2019 Sep;53(9):925-940. doi: 10.1111/medu.13914. Epub 2019 Jun 9. PMID 31179594
- [Background] Sewell JL, Bowen JL, Cate OT, O'Sullivan PS, Shah B, Boscardin CK. Learning Challenges, Teaching Strategies, and Cognitive Load: Insights From the Experience of Seasoned Endoscopy Teachers. Acad Med. 2020 May;95(5):794-802. doi: 10.1097/ACM.0000000000002946. PMID 31425188
- [Background] Kennedy TJ, Lingard LA. Making sense of grounded theory in medical education. Med Educ. 2006 Feb;40(2):101-8. doi: 10.1111/j.1365-2929.2005.02378.x. PMID 16451236
- See also: NASA-Task Load Index (TLX) scale — https://humansystems.arc.nasa.gov/groups/tlx/tlxpaperpencil.php
- See also: Joint Advisory Group on GI Endoscopy. Course Finder, JAG Endoscopy Training System — https://jetsapp.thejag.org.uk/courses
- See also: Canadian Association of Gastroenterology. Skills Enhancement for Endoscopy Program — https://www.cag-acg.org/education/see-program